CLINICAL TRIAL: NCT01179451
Title: Late Cardial Assessment in Children Who Were Diagnosed With Post Streptococcal Reactive Arthritis - a Long Term Study
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10040-10CTIL
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2012-03

CONDITIONS: Post Streptococcal Reactive Arthritis
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Post streptococcal reactive arthritis (PSRA): children who were diagnosed with psra at least one year before the study
  Interventions: Device: echocardiogram

INTERVENTIONS:
Device: echocardiogram — echocardiogram

SUMMARY:
The purpose of this study is to determine whether there is late cardial involvement in children diagnosed with post streptococcal reactive arthritis after discontinuation of prophylactic antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* PSRA patients under 18 who were diagnosed at least one year prior to the study

Exclusion Criteria:

* PSRA patients under 18 who were diagnosed less one year prior to the study
* patients who do not fulfill PSRA criteria
* patients who fulfill Jones criteria
* patients with a known heart defect

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: out patient rheumatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
cardiac valve function | at least 1 year after termination of antibiotic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel